CLINICAL TRIAL: NCT00277342
Title: Potential Association of a Common L-FABP Polymorphism With Lipid-induced Hepatic Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MOW_MM_LFABP
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2006-08

CONDITIONS: Wildtype; Polymorphism Liver FABP
Keywords: lipid induced hepatic insulin resistance; polymorphisms liver fatty-acid-binding-protein; gluconeogenesis; glycogenolysis; endogenous glucose production

INTERVENTIONS:
Procedure: measurement of lipid-induced hepatic insulin resistance

SUMMARY:
The investigators hypothesise that a common A277G polymorphism of the liver fatty acid binding protein (L-FABP) gene, which leads to an amino acid exchange, may be associated with alterations of lipid-induced hepatic insulin resistance. In the present study the investigators will investigate potential differences in lipid-induced hepatic insulin resistance, and in the relation between glycogenolysis and gluconeogenesis, in healthy subjects with the A277G polymorphism vs. subjects carrying the wildtype.

DETAILED DESCRIPTION:
Liver fatty acid binding protein (L-FABP) is an abundant cytosolic lipid-binding protein that regulates lipid transport and metabolism. Only one common non-synonymous polymorphism (A227G) leading to an amino-acid exchange in the exonic region of the L-FABP gene has been previously identified. Experimental elevations of free fatty acids (FFAs) have been shown to impair insulin mediated suppression of endogenous glucose production (EGP). Deletion of the L-FABP gene shows no obvious phenotype in mice receiving a low fat chow diet, but leads to decreased hepatic triglyceride accumulation in the prolonged fasted state, which exposes mice to an increased fatty acid flux to the liver. The function of the L-FABP gene may be altered by polymorphisms in coding regions of the gene, probably leading to modifications in hepatic triglyceride accumulation and hepatic insulin resistance.We hypothesize that carriers of the A277G SNP, when compared to matched wild-type subjects, may show altered responses of hepatic glucose production upon exposure to increased peripheral fatty acid concentrations, as achieved by lipid / heparin infusions. Because it is known that free fatty acids potently increase insulin secretion, we use somatostatin clamps in our experiments, followed by replacement of postabsorptive insulin and glucagon concentrations.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects with normal glucose tolerance (NGT)

Exclusion Criteria:

* any severe cardiac, liver, or kidney diseases
* pregnant or lactating women, menstrual irregularities
* cortisone, antidiabetic drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2006-01; Study Completion 2006-04

PRIMARY OUTCOMES:
lipid-induced hepatic insulin resistance(WT vs.SNP L-FABP)
changes in the relation GNG to GL

SECONDARY OUTCOMES:
changes in peripheral plasma glucose and lipid responses

CONTACTS AND LOCATIONS:
Overall Officials: Martin O Weickert, MD, Principal Investigator — German Institute of Human Nutrition; Charité Campus Benjamin Franklin; Matthias Möhlig, MD, Principal Investigator — German Institute of Human Nutrition; Charité Campus Benjamin Franklin; Andreas FH Pfeiffer, MD, Study Chair — German Institute of Human Nutrition; Charité Campus Benjamin Franklin
Locations (1):
- German Institute of Human Nutrition DIfE, Dpt. of Clinical Nutrition, Potsdam-Rehbrücke, Nuthetal, Germany

REFERENCES:
- [Result] Weickert MO, Loeffelholz CV, Roden M, Chandramouli V, Brehm A, Nowotny P, Osterhoff MA, Isken F, Spranger J, Landau BR, Pfeiffer AF, Mohlig M. A Thr94Ala mutation in human liver fatty acid-binding protein contributes to reduced hepatic glycogenolysis and blunted elevation of plasma glucose levels in lipid-exposed subjects. Am J Physiol Endocrinol Metab. 2007 Oct;293(4):E1078-84. doi: 10.1152/ajpendo.00337.2007. Epub 2007 Aug 14. PMID 17698986